CLINICAL TRIAL: NCT04265495
Title: Dual Trigger, Urinary HCG or Recombinant HCG, Which is the Best !? a Prospective Randomized Controlled Comparative Study
Brief Title: Dual Trigger, Urinary HCG or Recombinant HCG, Which is the Best !?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al Baraka Fertility Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, DOCTOR, Al Baraka Fertility Hospital
Other Study IDs: AlBarakaBH-KAMAL
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: IVF
Keywords: Dual trigger implantation,; HCG; OHSS; ANTAGONIST

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DUAL TRIGGERING: PATIENTS WILL RECEIVE DUAL TRIGGERING
- URINARY HCG: PATIENTS WILL RECEIVE URINARY HCG
- RECOMBINANT HCG: PATIENTS WILL RECEIVE RECOMBINANT HCG

SUMMARY:
a comparative study among dual trigger, urinary HCG and recombinant HCG regarding the outcome of ICSI- antagonist cycles

DETAILED DESCRIPTION:
a comparative study among dual trigger, urinary HCG and recombinant HCG regarding the outcome (oocyte quality, fertilization rate, implantation rate, clinical pregnancy rate as well as the incidence of OHSS) in ICSI- antagonist cycles

ELIGIBILITY:
Inclusion Criteria:

* patients <40 years of age who underwent IVF/ICSI cycles using a GnRH antagonist protocol

Exclusion Criteria:

* age: > 40 years
* BMI > 30 ,
* long agonist protocol
* were chromosomal and genetic disorders, abnormal ultrasonogram of the uterine cavity

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: patients <40 years of age who underwent IVF/ICSI cycles using a GnRH antagonist protocol, then at the time of triggering, we divided the patients to 3 groups by for triggering by a dual trigger, urinary HCG and recombinant HCG and then will check the outcome regarding the maturity and oocyte quality, implantation rate, clinical pregnancy rate as well as incidence of OHSS
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate, | 4 WEEKS
implantation rate, | 2 WEEKS
incidence of OHSS. | 1 WEEK

CONTACTS AND LOCATIONS:
Locations (1):
- Al-BARAKA FERTILITY HOSPITAL, Manama, Adliya, Bahrain